CLINICAL TRIAL: NCT01860976
Title: A Phase 3 Randomized Placebo-Controlled Study to Evaluate the Efficacy and Safety of Abatacept Subcutaneous Injection in Adults With Active Psoriatic Arthritis
Brief Title: Efficacy and Safety of Subcutaneous Abatacept in Adults With Active Psoriatic Arthritis
Acronym: ASTRAEA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM101-332; 2012-002798-80 (EudraCT Number)
Record Dates: First submitted 2013-05-21; First posted 2013-05-23 (Estimated); Results first posted 2017-08-02 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Abatacept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Abatacept (Experimental): Abatacept 125 mg/syringe (125 mg/mL) solution subcutaneously once a week for 168 days double blind/197 days open label/365 days long term extension
  Interventions: Drug: Abatacept
- Placebo (Placebo Comparator): Placebo matching with Abatacept 0 mg solution subcutaneously once a week 168 days double blind
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Abatacept
  Other Names: Orencia
  Arms: Abatacept
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare subcutaneous Abatacept to placebo in the treatment of psoriatic arthritis

DETAILED DESCRIPTION:
ASTRAEA=Active PSoriaTic ARthritis RAndomizEd TriAl

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Subjects at least 18 years of age who have a diagnosis of PsA by Classification Criteria for Psoriatic Arthritis (CASPAR)
* Subjects have active PsA as shown by a minimum of ≥3 swollen joints and ≥3 tender joints (66/68 joint counts) at screening and randomization/Day 1 (prior to study drug administration). At least one of the swollen joints must be in the digit of the hand or foot
* Subjects with at least one confirmed ≥2 cm target lesion of plaque psoriasis in a region of the body that can be evaluated excluding the axilla, genitals, groin, palms, and soles
* Subjects must have had an inadequate response or intolerance to at least one non-biologic disease-modifying anti-rheumatic drug (DMARD)
* Subjects may have been exposed to TNFi therapy. Subjects may have discontinued for any reason (inadequate response, intolerance or other)
* Subjects may enroll on certain concomitant non-biologic DMARDs (Methotrexate, Leflunomide, Sulfasalazine, or Hydroxychloroquine) provided the medication has been used for at least 3 months with a stable dose for at least 28 days prior to randomization (Day 1)
* If using oral corticosteroids (≤10 mg mg/day Prednisone equivalent), dose must be stable ≥14 days prior to randomization (Day 1)
* Subjects may enroll on systemic retinoids (eg: Acitretin) provided the medication has been used for at least 3 months with a stable dose for at least 28 days prior to randomization (Day 1)

Exclusion Criteria:

* Subjects with guttate, pustular, or erythrodermic psoriasis
* Subjects who have had prior exposure to Abatacept (CTLA 4Ig) or other CTLA4 therapies
* Subjects who have been exposed to any investigational drug within 4 weeks or 5 half lives, whichever is longer
* Female subjects who had a breast cancer screening study that is suspicious for malignancy, and in whom the possibility of malignancy cannot be reasonably excluded following additional clinical, laboratory or other diagnostic evaluations
* Subjects with a history of cancer within the last 5 years (other than non-melanoma skin cell cancers cured by local resection). Existing non-melanoma skin cell cancers must be removed prior to dosing. Subjects with carcinoma in situ, treated with definitive surgical intervention prior to study enrollment are allowed
* Subjects with any bacterial infection within the last 60 days prior to screening (enrollment), unless treated and resolved with antibiotics, or any chronic bacterial infection (such as chronic pyelonephritis, osteomyelitis and bronchiectasis)
* Subjects at risk for tuberculosis (TB). Specifically, subjects with:

  * Current clinical, radiographic or laboratory evidence of active TB
  * A history of active TB within the last 3 years even if it was treated
  * A history of active TB greater than 3 years ago unless there is documentation that the prior anti-TB treatment was appropriate in duration and type
  * Latent TB which was not successfully treated
  * Subjects with a positive TB screening test indicative of latent TB will not be eligible for the study unless they have no evidence of current TB on chest x-ray at screening and they are actively being treated for TB with isoniazid (INH) or other therapy for latent TB given according to local health authority guidelines (eg: Center for Disease Control). Treatment must have been given for at least 4 weeks prior to randomization (Day 1). These subjects should complete treatment according to local health authority guidelines
* Subjects with herpes zoster that resolved less than 2 months prior to enrollment
* Subjects with evidence (as measured by the investigator) of active or latent bacterial, active viral, or serious latent viral infections at the time of enrollment, including subjects with evidence of Immunodeficiency Virus (HIV) infection
* Subjects who are not currently treated with a non-biologic DMARD and have clinical or radiographic evidence of arthritis mutilans (eg: digital telescoping or "pencil-in-cup" radiographic changes)
* Subjects who have failed more than 2 TNFi due to inefficacy defined as inadequate response after 3 months treatment at a therapeutic dose
* Subjects who have received TNFi therapy within 4 weeks for etanercept or within 8 weeks for adalimumab, certolizumab, infliximab, or golimumab
* Subjects who have received prior use of apremilast within 4 weeks, ustekinumab within 20 weeks or briakinumab within 8 weeks
* Subjects who have discontinued a non-biologic DMARD or systemic retinoid within four weeks or five half-lives, whichever is longer, prior to randomization (Day 1)
* Use of any of the following within 28 days or five half lives whichever is longer prior to randomization (Day 1): Cyclosporine A, oral Tacrolimus, Mycophenolate Mofetil (MMF), Hydroxyurea, Fumaric Acid Esters, Paclitaxel, 6-Thioguanine, 6-Mercatopurine, or Tofacitinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 489 (Actual)
Dates: Start 2013-06-17 (Actual); Primary Completion 2015-07-14 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (78):
- United States (17):
  - Arizona Arthritis & Rheumatology Research PLLC, Phoenix, Arizona
  - Arthritis Asso & Osteo Ctr Of Colorado Springs, Colorado Springs, Colorado
  - Joao Nascimento, Bridgeport, Connecticut
  - New England Research Associates, Llc, Trumbull, Connecticut
  - Sarasota Arthritis Research Center, Sarasota, Florida
  - Klein And Associates, M.D., Pa, Hagerstown, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - St. Paul Rheumatology, P.A., Eagan, Minnesota
  - Box Arthritis And Rheumatology Of The Carolinas, Pllc, Charlotte, North Carolina
  - Paramount Medical Research & Consulting, Llc, Middleburg Heights, Ohio
  - Health Research Of Oklahoma, Oklahoma City, Oklahoma
  - East Penn Rheumatology Associates, P.C., Bethlehem, Pennsylvania
  - Clinical Research Center Of Reading, Llc, Wyomissing, Pennsylvania
  - West Tennessee Research Institute, Jackson, Tennessee
  - Rheumatology Consultants Pllc, Knoxville, Tennessee
  - Seattle Rheumatology Associates, Seattle, Washington
  - Arthritis Northwest, Spokane, Washington
- Argentina (6):
  - Local Institution, Ciudad Autonoma Beunos Aires, Buenos Aires
  - Instituto de Asistencia Reumatologica Integral, San Fernando, Buenos Aires
  - Caici, Rosario, Santa Fe Province
  - Centro Medico Privado De Reumatologia, San Miguel de Tucumán, Tucumán Province
  - Instituto De Rehabilitacion Psicofisica, Buenos Aires
  - Instituto Reumatologico Strusberg, Córdoba
- Brazil (2):
  - Local Institution, Juiz de Fora, Minas Gerais
  - Local Institution, Curitiba, Paraná
- Canada (4):
  - Nexus Clinical Research, St. John's, Newfoundland and Labrador
  - Toronto Western Hospital, University Health Network, Toronto, Ontario
  - Manna Research, Toronto, Ontario
  - Groupe De Recherche En Rhumatologie Et Maladies Osseuses, Québec, Quebec
- Chile (3):
  - Local Institution, Viña del Mar, Región de Valparaíso
  - Local Institution, Santiago, Santiago Metropolitan
  - Local Institution, Santiago
- Colombia (3):
  - Riesgo De Fractura, Bogota, Cundinamarca
  - Servimed E.U, Bucaramanga
  - Clinica de Artritis Temprana, Cali
- Local Institution, Prague, Czechia
- France (5):
  - Local Institution, Chambray-lès-Tours
  - Local Institution, Lille
  - Local Institution, Montpellier
  - Local Institution, Poitiers
  - Local Institution, Strasbourg
- Germany (7):
  - Local Institution, Bad Abbach
  - Local Institution, Erlangen
  - Local Institution, Freiburg im Breisgau
  - Local Institution, Hamburg
  - Local Institution, München
  - Local Institution, Ratingen
  - Local Institution, Trier
- Greece (2):
  - Local Institution, Athens
  - Local Institution, Crete
- Israel (4):
  - Local Institution, Ashkelon
  - Local Institution, Haifa
  - Local Institution, Ramat Gan
  - Local Institution, Tel Aviv
- Italy (4):
  - Local Institution, Florence
  - Local Institution, Milan
  - Local Institution, Palermo
  - Local Institution, Viale Europa Cantanzaro
- Mexico (6):
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Zapopan, Jalisco
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Monterrey, N.l., Nuevo León
  - Local Institution, Mérida, Yucatán
  - Local Institution, Aguascalientes
- Peru (3):
  - Clinica San Felipe, Lima
  - Hospital Nacional Guillermo Almenara Irigoyen, Lima
  - Instituto De Ginecologia Y Reproduccion Inv. Clinical Sac, Lima
- Poland (4):
  - Local Institution, Elblag, Warminsko-mazurski
  - Local Institution, Dąbrówka
  - Local Institution, Mysłowice
  - Local Institution, Warsaw
- South Africa (4):
  - Local Institution, Pretoria, Gauteng
  - Local Institution, Cape Town, Western Cape
  - Local Institution, Pinelands, Cape Town, Western Cape
  - Local Institution, Stellenbosch, Western Cape
- Spain (3):
  - Local Institution, A Coruña
  - Local Institution, Santander
  - Local Institution, Seville

REFERENCES:
- [Derived] McInnes IB, Ferraccioli G, D'Agostino MA, Le Bars M, Banerjee S, Ahmad HA, Elbez Y, Mease PJ. Body mass index and treatment response to subcutaneous abatacept in patients with psoriatic arthritis: a post hoc analysis of a phase III trial. RMD Open. 2019 May 30;5(1):e000934. doi: 10.1136/rmdopen-2019-000934. eCollection 2019. PMID 31245054
- [Derived] Strand V, Alemao E, Lehman T, Johnsen A, Banerjee S, Ahmad HA, Mease PJ. Improved patient-reported outcomes in patients with psoriatic arthritis treated with abatacept: results from a phase 3 trial. Arthritis Res Ther. 2018 Dec 6;20(1):269. doi: 10.1186/s13075-018-1769-7. PMID 30522501
- [Derived] Mease PJ, Gottlieb AB, van der Heijde D, FitzGerald O, Johnsen A, Nys M, Banerjee S, Gladman DD. Efficacy and safety of abatacept, a T-cell modulator, in a randomised, double-blind, placebo-controlled, phase III study in psoriatic arthritis. Ann Rheum Dis. 2017 Sep;76(9):1550-1558. doi: 10.1136/annrheumdis-2016-210724. Epub 2017 May 4. PMID 28473423
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 424 were Randomized and Treated
Groups:
- Abatacept: Abatacept 125mg, self-administered subcutaneously, once weekly
- Placebo: Placebo, self-administered subcutaneously, once weekly.
Period: Blinded Treatment
Arm/Group | Abatacept | Placebo
Started | 213 | 211
Completed (completed = participants who completed treatment period) | 125 | 98
Not Completed | 88 | 113
Not completed — Adverse Event | 1 | 3
Not completed — Lack of Efficacy | 5 | 12
Not completed — Subject request to discontinue treatment | 2 | 3
Not completed — Withdrawal by Subject | 3 | 5
Not completed — Subject no longer met criteria | 1 | 0
Not completed — Entered Open-Label in error | 0 | 1
Not completed — Early Escape: Transitioned to OL period | 76 | 89
Period: Open-Label
Arm/Group | Abatacept | Placebo
Started | 197 | 185
Completed (completed = participants who completed the open label period) | 169 | 166
Not Completed | 28 | 19
Not completed — Adverse Event | 2 | 4
Not completed — Lack of Efficacy | 16 | 8
Not completed — Lost to Follow-up | 1 | 2
Not completed — Subject request discontinue treatment | 4 | 3
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Other Reasons | 1 | 1
Period: Long Term Extension
Arm/Group | Abatacept | Placebo
Started | 106 | 0
Completed (completed = completed long term extension period at the time of analysis) | 81 | 0
Not Completed | 25 | 0
Not completed — Adverse Event | 4 | 0
Not completed — Lack of Efficacy | 2 | 0
Not completed — Subject request to discontinue treatment | 10 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — subject withdrew consent | 7 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Abatacept | Placebo | Total
Number analyzed (Participants) | 213 | 211 | 424
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.0 (10.67) | 49.8 (11.26) | 50.4 (10.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121 | 112 | 233
  Male | 92 | 99 | 191
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 195 | 198 | 393
  More than one race | 18 | 11 | 29
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of ACR 20 Responders at Day 169
Description: The American College of Rheumatology (ACR) 20 definition of improvement is a 20% improvement over baseline in tender and swollen joint counts and a 20% improvement in 3 of the 5 remaining core data set measures (participant global assessment of pain, participant global assessment of disease activity, physician global assessment of disease activity, participant assessment of physical function, acute phase reactant value). The number of ACR 20 responders was divided by the number of treated participants and expressed as a percentage. Early escape participants, and participants with missing data at day 169 were imputed as non-responders.
Time Frame: Day 169
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 213 | 211
Percentage of participants | 39.4 [32.9 to 46.0] | 22.3 [16.7 to 27.9]
Statistical Analysis 1: Comparison: Abatacept vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Estimate of Difference = 17.2, 95% CI 2-sided [8.7 to 25.6]

2. Secondary Outcome: Proportion of Health Assessment Questionnaire (HAQ) Responders at Day 169
Description: Participants were considered responders if their HAQ score decreased at least 0.35 from baseline. The number of HAQ responders was divided by the number of treated participants and expressed as a percentage. Scoring conventions are based on the Standard Disability Index of HAQ/HAQ-DI using the 20 response items. For each of the 8 disability categories there is an "aids/devices" companion variable that is used to record the type of assistance, if any, a participant uses for his/her usual activities. If either "aids/devices" and/or "assistance from another person" are checked for a disability category, the score for this category is set to "2" (much difficulty), if the original score was "0" (no difficulty) or "1" (some difficulty). The HAQ-DI is then calculated by summing the adjusted categories scores and dividing by the number of categories answered. Early escape participants, and participants with missing data at day 169 were imputed as non-responders.
Time Frame: Baseline to Day 169
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 213 | 211
percentage of participants | 31.0 [24.8 to 37.2] | 23.7 [18.0 to 29.4]

3. Secondary Outcome: Proportion of ACR 20 Responders at Day 169 in the TNFi-naïve Subpopulation
Description: The ACR 20 definition of improvement is a 20% improvement over baseline in tender and swollen joint counts and a 20% in 3 of the 5 remaining core data set measures (participant global assessment of pain, participant global assessment of disease activity, physician global assessment of disease activity, participant assessment of physical function, acute phase reactant value). The number of ACR 20 responders was divided by the number of treated, TNFi-naive participants and expressed as a percentage. Early escape participants, and participants with missing data at day 169 were imputed as non-responders.
Time Frame: Day 169
Population: All treated TNFi-naïve participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 84 | 81
Percentage of participants | 44.0 [33.4 to 54.7] | 22.2 [13.2 to 31.3]

4. Secondary Outcome: Proportion of ACR 20 Responders at Day 169 in the TNFi-exposed Subpopulation
Description: The ACR 20 definition of improvement is a 20% improvement over baseline in tender and swollen joint counts and a 20% in 3 of the 5 remaining core data set measures (participant global assessment of pain, participant global assessment of disease activity, physician global assessment of disease activity, participant assessment of physical function, acute phase reactant value). The number of ACR 20 responders was divided by the number of treated, TNFi-exposed participants and expressed as a percentage. Early escape participants, and participants with missing data at day 169 were imputed as non-responders.
Time Frame: Day 169
Population: All treated TNFi-exposed participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 129 | 130
Percentage of participants | 36.4 [28.1 to 44.7] | 22.3 [15.2 to 29.5]

5. Secondary Outcome: Proportion of Non-progressors in Total PsA-modified SHS at Day 169
Description: The number of radiographic non-progressors in total PsA-Modified Sharp van der Heijde score (SHS) at Day 169 was divided by the number of treated participants and expressed as a percentage. Non-progression was defined as a change from baseline in total PsA modified SHS ≤0. Early escape participants, and participants with missing data at day 169 were imputed as non-progressors.
Time Frame: Baseline to Day 169
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 213 | 211
Percentage of participants | 42.7 [36.1 to 49.4] | 32.7 [26.4 to 39.0]

6. Secondary Outcome: Proportion of Participants Achieving a PASI 50 at Day 169 in Participants With Baseline BSA >= 3%
Description: The number of participants who achieved at least 50% improvement from baseline in Psoriasis Area and Severity Index Arthritis (PASI 50) at Day 169 was divided by the number of treated participants with BSA >= 3% and expressed as a percentage. Only participants with >= 3% body surface area (BSA) of psoriatic skin involvement at randomization were included in this analysis.
Time Frame: Baseline to Day 169
Population: All treated participants with >= 3% BSA of psoriatic skin involvement at randomization
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 146 | 148
Percentage of participants | 26.7 [19.5 to 33.9] | 19.6 [13.2 to 26.0]

7. Secondary Outcome: Proportions of ACR 50 and ACR 70 Responders at Day 169
Description: The ACR 50 and ACR 70 definition of improvement is a 50% or 70% improvement, respectively, over baseline in tender and swollen joint counts and a 50% or 70% improvement in 3 of the 5 remaining core data set measures (participant global assessment of pain, participant global assessment of disease activity, physician global assessment of disease activity, participant assessment of physical function, acute phase reactant value). The number of ACR 50 and ACR 70 responders was divided by the number of treated participants and expressed as a percentage. Early escape participants, and participants with missing data at day 169 were imputed as non-responders.
Time Frame: Day 169
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 213 | 211
Percentage of participants
  ACR 50 | 19.2 [14.0 to 24.5] | 12.3 [7.9 to 16.8]
  ACR 70 | 10.3 [6.2 to 14.4] | 6.6 [3.3 to 10.0]

8. Secondary Outcome: Mean Change From Baseline in SF-36 Physical and Mental Components at Day 169
Description: Adjusted mean change in scores on the Short Form 36 physical and mental function assessment (SF-36) from baseline were analyzed from the physical component summary (PCS) mental component summary (MCS). The SF-36 is a participant questionnaire assessing 8 domains of health status: physical functioning, pain, vitality, social functioning, psychological functioning, general health perception, and role limitations due to physical and emotional problems. The instrument can be divided into two summary scores, physical and mental component score. The scores range from 0 to 100, with a higher score indicating better quality of life. The two summary scores (PCS and MCS) will be calculated by taking a weighted linear combination of the 8 individual subscales.
Time Frame: Baseline to Day 169
Population: All treated participants
Measure: Mean (Standard Error); unit: SF-36 points
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 213 | 211
SF-36 points
  PCS | 5.11 (0.637) | 3.69 (0.707)
  MCS | 2.56 (0.826) | 2.62 (0.924)

9. Secondary Outcome: Proportion of Participants With at Least One Positive Immunogenicity Response up to Day 169 Relative to Baseline
Description: Blood samples were collected at Days 1, 85 and 169 and assayed for the presence of abatacept-specific antibodies. The number of participants with at least one positive immunogenicity response was divided by the number of treated participants and expressed as a percentage.
Time Frame: Baseline to Day 169
Population: All treated participants
Measure: Number; unit: Percentage of participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 203 | 198
Percentage of participants | 3.9 | 8.6

10. Secondary Outcome: Proportion of Participants With AEs at Day 169
Description: Proportion of participants with AEs at Day 169
Time Frame: Day 169
Population: All Treated Participants
Measure: Number; unit: Percentage of participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 213 | 211
Percentage of participants | 54.5 | 53.1

11. Secondary Outcome: Proportion of Participants With SAEs at Day 169
Description: Proportion of participants with SAEs at Day 169
Time Frame: Day 169
Population: All Treated Participants
Measure: Number; unit: Percentage of participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 213 | 211
Percentage of participants | 2.8 | 4.3

12. Secondary Outcome: Proportion of Participants With AEs Leading to Discontinuation at Day 169
Description: Proportion of participants with AEs leading to discontinuation at Day 169
Time Frame: Day 169
Population: All Treated Participants
Measure: Number; unit: Percentage of participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 213 | 211
Percentage of participants | 1.4 | 1.9

13. Secondary Outcome: Proportion of Participant Deaths at Day 169
Description: Proportion of participant deaths at Day 169
Time Frame: Day 169
Population: All Treated Participants
Measure: Number; unit: Percentage of participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 213 | 211
Percentage of participants | 0 | 0

14. Secondary Outcome: Proportion of Participants With Marked Laboratory Abnormalities at Day 169
Description: Proportion of participants with marked laboratory abnormalities at Day 169
Time Frame: Day 169
Population: All Treated Participants
Measure: Number; unit: Percentage of participants
Arm/Group | Abatacept | Placebo
Number analyzed (Participants) | 213 | 211
Percentage of participants | 3.2 | 5.4

ADVERSE EVENTS:
Time Frame: Up to 56 days post last dose in the short-term period or the first dose in the open-label period, whichever occurs first
Arm/Group | ABATACEPT DURING DOUBLE-BLIND PERIOD | PLACEBO DURING DOUBLE-BLIND PERIOD | ABATACEPT DURING OPEN-LABEL PERIOD | ABATACEPT DURING OPEN-LABEL EXTENSION PERIOD | ABATACEPT DURING LONG-TERM EXTENSION PERIOD
All-Cause Mortality (participants affected / at risk) | 0/213 | 0/211 | 0/382 | 0/322 | 0/106
Serious Adverse Events (participants affected / at risk) | 6/213 | 9/211 | 29/382 | 20/322 | 17/106
Other Adverse Events (participants affected / at risk) | 39/213 | 43/211 | 92/382 | 103/322 | 56/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABATACEPT DURING DOUBLE-BLIND PERIOD (N=213) | PLACEBO DURING DOUBLE-BLIND PERIOD (N=211) | ABATACEPT DURING OPEN-LABEL PERIOD (N=382) | ABATACEPT DURING OPEN-LABEL EXTENSION PERIOD (N=322) | ABATACEPT DURING LONG-TERM EXTENSION PERIOD (N=106)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Dermoid cyst (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0
Meniere's disease (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastric mucosa erythema (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0
Incarcerated hernia (General disorders) | 0 | 0 | 1 | 0 | 0
Biliary dilatation (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 1 | 1 | 1
Hepatic fibrosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Epstein-Barr virus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 0 | 0 | 0 | 1
Groin abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Intervertebral discitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumocystis jirovecii infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 4 | 2
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 3 | 3
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Carcinoma in situ of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Demyelination (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Calculus bladder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Polycystic ovaries (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Acute chest syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Erythrodermic psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Peripheral artery thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Venous thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ABATACEPT DURING DOUBLE-BLIND PERIOD (N=213) | PLACEBO DURING DOUBLE-BLIND PERIOD (N=211) | ABATACEPT DURING OPEN-LABEL PERIOD (N=382) | ABATACEPT DURING OPEN-LABEL EXTENSION PERIOD (N=322) | ABATACEPT DURING LONG-TERM EXTENSION PERIOD (N=106)
Bronchitis (Infections and infestations) | 7 | 5 | 19 | 17 | 15
Influenza (Infections and infestations) | 4 | 3 | 9 | 17 | 4
Nasopharyngitis (Infections and infestations) | 9 | 11 | 17 | 26 | 16
Pharyngitis (Infections and infestations) | 0 | 2 | 5 | 10 | 6
Upper respiratory tract infection (Infections and infestations) | 6 | 14 | 23 | 19 | 3
Urinary tract infection (Infections and infestations) | 10 | 2 | 10 | 12 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 10 | 11 | 12
Sciatica (Nervous system disorders) | 1 | 0 | 2 | 1 | 6
Catarrh (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2 | 12
Hypertension (Vascular disorders) | 5 | 8 | 10 | 7 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-08-19): https://cdn.clinicaltrials.gov/large-docs/76/NCT01860976/Prot_SAP_000.pdf